CLINICAL TRIAL: NCT02183766
Title: Effect of the Prebiotic 4'Galactooligosaccharides in Children and Adolescents With Functional Constipation
Brief Title: GOS Prebiotic Effect in Children Constipation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Celia Aparecida Valbon Beleli, Master, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 366/2009; 0280.0.146.000-09 (Other: CAAE)
Record Dates: First submitted 2014-06-26; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maltodextrin (Placebo Comparator): 6 mL once a day diluted in juice during 30 days.
  Interventions: Drug: Maltodextrin
- Galactooligosaccharide prebiotic (Active Comparator): 6 mL once a day diluted in juice during 30 days.
  Interventions: Dietary Supplement: Galactooligosaccharide prebiotic

INTERVENTIONS:
Dietary Supplement: Galactooligosaccharide prebiotic — 6 mL once a day
  Arms: Galactooligosaccharide prebiotic
Drug: Maltodextrin — 6 mL once a day
  Other Names: Placebo
  Arms: Maltodextrin

SUMMARY:
Some prebiotics are useful for improving symptoms related to constipation, but clinical trials including infants and older children are scarce. A double-blind, placebo-controlled, crossover clinical trial was conducted to evaluate the effect of galactooligosaccharides (GOS) on functional constipation in children and adolescents. Twenty children aged 4 to 16 years of age, who spontaneously sought medical care at a primary healthcare unit, received 1.7g GOS or placebo (Maltodextrin) treatment for 30 days, followed by a 15-day washout period and a 30-day use of an alternative product. A clinical score was calculated at baseline, at the 15th (D15) and 30th (D30) day of each period, to assess bowel movement frequency, straining/ pain during defecation and stool consistency. Oral anal transit time with activated charcoal was determined at baseline and D30 of each period.

DETAILED DESCRIPTION:
Constipation is a common symptom in the pediatric clinics. It is usually defined in terms of difficulty of passage of faeces, faecal consistency and frequency of evacuation. A diet containing high amounts in fiber can promote beneficial effects constipation therapy. Beside the fiber, functional foods, such as prebiotics, have been considered useful to regulate bowel movements. Prebiotic is defined as nondigestible food components that affect the host for stimulating selectively growth of potentially beneficial bacteria in the intestines, specially the colon. Nowadays, there are few clinical trials evaluating prebiotic use for relieving constipation symptoms in children. This clinical trial aimed to evaluate the effect of Galactooligossacharides (GOS) on constipated children. The trial consisted of a 75-day period double blind intervention, controlled with placebo and cross over delimitation, with two sequences of evaluation and two treatments, placebo and galactooligossacharides. It included 20 children (4-16 years) with functional constipation defined by the ROMA III criteria. Children have received 6g of GOS or 6g Maltodextrin (placebo), the solution was ingested for 30 days, followed by a washout period of 15 days, and afterwards, 30 more days of GOS or Maltodextrin, alternately with the product ingested in the first 30 days. The study was designed according to crossover delimitation (GOS and Placebo). Eleven patients were evaluated according to the sequence GOS/placebo and nine patients with the sequence Placebo/GOS. A severity score was measured at the beginning, 2nd and 4th week in each experiment. Clinical scores, elaborated for this Trial, were used to evaluate the effect of the products considering: stool frequency, presence of pain/discomfort/effort during evacuation, consistency of stool and loss of appetite or early satiety. Scores were calculated at day zero (D0), 15th day (D15) and 30th day (D30) of the study, in each phase of the "crossover". Oroanal transit evaluation was performed on D0 and D30 of each sequence, by activated charcoal ingestion.

Descriptive analysis trough measures of position and dispersion were realized for numerical variables. ANOVA was used for the analysis of GOS effect. The significance level assumed for the statistical tests was 5%. The GOS presented significant effect compared to placebo, reducing the stool consistency p< 0,0001 and rising the stool frequency, p=0,0014. The value of the oroanal transit time were significant lower in GOS period, p<0,0001. GOS was effective at the improvement of mild constipation symptoms and may represent an alternative option for the therapy of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Functional constipation defined by Rome III criteria
* Consent form signed by parent or guardian

Exclusion Criteria:

* Patients with systemic, genetic or neurological diseases.
* Lactose intolerance
* Laxative use
* Probiotic use
* Antibiotic use during the study

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evidence of constipation improvement after GOS use in children compared to use of placebo. | within 30 days of GOS use.

CONTACTS AND LOCATIONS:
Overall Officials: Celia Beleli, Master, Principal Investigator — University of Campinas